CLINICAL TRIAL: NCT05429749
Title: Intravenous Iron Supplement to Prevent Postoperative Delirium After Hip Fracture Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: JW Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Young-Kyun Lee, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ferinject
Record Dates: First submitted 2022-04-17; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ferinject group (Experimental): This group of hip fracture patients are treated with intravenous Ferinject between the admission and the surgery day.
  Interventions: Drug: Ferinject
- Control group (Active Comparator): This group of hip fracture patients are treated with normal saline as a control group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ferinject — Intravenous ferinject 1000mg is administered between the admission day and the surgery day.
  Other Names: Ferric Carboxymaltose
  Arms: Ferinject group
Drug: Normal saline — Normal saline 250ml is administered between the admission day and the surgery day.
  Arms: Control group

SUMMARY:
This is a clinical trial to evaluate the effect of intravenous iron supplement with Ferinject (Ferric Carboxymaltose) in preventing postoperative delirium after hip fracture surgery.

DETAILED DESCRIPTION:
We hypothesized that IV iron supplement will (1) decrease postoperative delirium in hip fracture patients and (2) decrease the amount of transfusion and transfusion-related complications.

ELIGIBILITY:
Inclusion Criteria:

* femur neck fracture, intertrochanteric fractures
* Iron deficiency anemia (Hb<12 in women, Hb<13 in men)
* Iron deficiency (Serum ferritin <100ug/L or transferrin saturation<20%)
* Who understands this clinical trial and volunteers and agrees to this trial

Exclusion Criteria:

* Patient under the age of 65 years
* Hb<7 or someone who has acute symptom of anemia(tachycardia, dyspnea, or dizziness)
* High energy trauma
* Preoperative delirium
* MMSE<10
* Underlying disease which involves cognitive dysfunction (e.g. neurovascular diseases, acute myocardial infarction, pulmonary embolism)
* Those who are inappropriate to participate in the clinical trial assessed by the investigators

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium | since immediately after the surgery to the discharge date
  The presence and duration of postoperative delirium

SECONDARY OUTCOMES:
Postoperative transfusion | Postoperative admission datessince immediately after the surgery to the discharge date
  The amount of postoperative transfusion
Transfusion-related complications | since immediately after the surgery to the discharge date
  The presence of transfusion-related complications
Functional outcomes | since immediately after the surgery to the discharge date
  Postoperative functional outcomes of hip fracture patients
Hematologic outcomes | since immediately after the surgery to the discharge date
  Postoperative hematologic outcomes of hip fracture patients

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea